CLINICAL TRIAL: NCT04849000
Title: Phase III, Multicentre, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Efficacy and Safety of SHR-1209 Monotherapy in Patients With Primary Hypercholesterolemia and Mixed Hyperlipemia
Brief Title: Study of SHR-1209 in the Treatment of Hypercholesterolemia and Hyperlipidemia Ⅲ Stage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1209-301
Record Dates: First submitted 2021-03-31; First posted 2021-04-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-06

CONDITIONS: Primary Hypercholesterolemia; Mixed Hyperlipemia
MeSH Terms: conditions — Hyperlipoproteinemia Type V

STUDY DESIGN:
Intervention Model Description: SHR-1209 monotherapy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1209 (Experimental)
  Interventions: Drug: SHR-1209
- SHR-1209 Placebo (Placebo Comparator)
  Interventions: Drug: SHR-1209 Placebo

INTERVENTIONS:
Drug: SHR-1209 — SHR-1209
  Arms: SHR-1209
Drug: SHR-1209 Placebo — SHR-1209 Placebo
  Arms: SHR-1209 Placebo

SUMMARY:
The study is ongoing to evaluate the efficacy and safety of SHR-1209 in patients with hypercholesterolemia and hyperlipemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤80 on the date of signing the informed consent, male or female;
2. Fasting LDL-C was ≥2.6mmol/L and <4.9mmol/L at screening and randomization；
3. Those who understand the study procedures and methods, volunteer to participate in the study, and sign the informed consent in person.

Exclusion Criteria:

1. Have the following diseases or treatment history :(1) Have known allergic reaction to experimental drugs, or have severe allergic reaction to other antibody drugs;(2) previous diagnosis of cardiac function as defined by the New York Heart Association (NYHA) grade III-IV;
2. Any of the laboratory indicators met the following criteria at screening or at random :(1) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding 2 times the upper limit of normal (ULN), or total bilirubin exceeding 1.5 times the upper limit of normal (ULN);(2) Creatine kinase (CK) exceeds 3 times the upper limit of normal value (ULN);
3. General conditions :(1) the investigator judged that subcutaneous injection was not appropriate;(2) Fertile female subjects who did not use contraception within 4 weeks before screening;Or male or female subjects who do not agree to use high-efficiency contraceptives during the trial and for 24 weeks after the last dosing;(3) Women who are pregnant or lactating.
4. The Investigator determines that the subjects have poor compliance or have any factors that may prevent them from participating in the study, including, but not limited to, the study placing the subjects at unacceptable risk or possibly interfering with the study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
12-weeks or 16weeks Percentage change in LDL-C relative to baseline | 12-weeks or 16weeks

SECONDARY OUTCOMES:
12-weeks or 16weeks change in LDL-C relative to baseline； | 12-weeks or 16weeks
Percentage of changes in non-HDL-C, ApoB, TC/HDL-C, ApoB/ApoA1, LP (a) and TG relative to baseline and relative to baseline after 12 weeks or 16 weeks of treatment | 12 weeks or 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangzhou, China

REFERENCES:
- [Derived] Shu C, Wang Y, Feng S, Yang S, Shen K. Population Pharmacokinetics and Pharmacodynamics Modeling for the Use of Recaticimab in Healthy Volunteers and Patients with Hypercholesterolemia. Clin Pharmacokinet. 2025 Sep;64(9):1341-1355. doi: 10.1007/s40262-025-01512-5. Epub 2025 Jun 30. PMID 40587053